CLINICAL TRIAL: NCT02539615
Title: A Single-arm, Multi-center Trial of the ForeCYTE Breast Aspirator for Sample Collection and Cytological Testing of Nipple Aspirate Fluid in Women 30-55 Years of Age
Brief Title: A Trial of the ForeCYTE Breast Aspirator for Cytological Testing of Nipple Aspirate Fluid in Women 30-55 Years Old
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Atossa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GCP005
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer, Preneoplastic Conditions, BRCA
MeSH Terms: conditions — Breast Neoplasms; Precancerous Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ForeCYTE Breast Aspirator - Nipple Aspirate Fluid Collection (Experimental): Nipple Aspirate is collected using the ForeCYTE Breast Aspirator
  Interventions: Device: ForeCYTE Breast Aspirator

INTERVENTIONS:
Device: ForeCYTE Breast Aspirator

SUMMARY:
The purpose of this study is to measure the performance of the ForeCYTE Breast Aspirator for the collection and processing of Nipple Aspirate Fluid (NAF) specimens for cytology. Including collecting, processing and shipping samples, training staff, processing samples, sample interpretation and accurate and timely reporting in a manner resembling routine clinical use. The study will include a subset of patients who are known carriers of a BRCA germline mutation. NAF from this subset will be submitted for molecular testing in addition to cytology.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, female, age 30-55 years, from whom bi-lateral specimens can be obtained.

   The following additional considerations apply:
   * Women with prior mastectomy/lumpectomy may be considered for NAF-collection in the contralateral (non-operated) breast only if they were:

     * Stage I or Stage II at the time of surgery;
     * Have completed any and all hormonal therapy, chemotherapy, or targeted therapy at least one year prior to inclusion;
     * Are considered disease-free (NED- No Evidence of Disease) at the time of study entry;
   * Women under the age 30 may be enrolled if they are within 10 years of the age at diagnosis of breast cancer in a first-degree relative. No subject under the age of 21 may be enrolled.
2. Any woman for whom NAF-cytology testing is considered to be beneficial by her physician. This includes, but is not limited to women with first- and/or second degree relatives with breast- or ovarian cancer. Known presence of a BRCA-1 or BRCA-2 germline mutation is allowed but not required. If known, any such mutation will be noted on the Case Report Form. The protocol does not provide for testing of women without known germ-line mutations.
3. Non-lactating and non-pregnant.
4. Good general health as determined by medical history, breast disease/cancer history, and clinical breast exam.
5. Willing to give informed consent and follow study procedures as directed.

Exclusion Criteria

1. Medical condition/psychiatric conditions making subjects a poor candidate for study, as determined by the Principal Investigator.
2. Pregnancy or suspicion of pregnancy.
3. Open cutaneous wounds or atopic dermatitis in the area of the nipple-areolar complex.
4. No or inverted nipple on the breast unfit for fluid collection, or significant prior surgery in the area of the nipple-areolar complex.
5. Participation in an investigational drug or device study less than 30 days prior to enrollment in this study.
6. Pregnancy, childbirth, or lactation less than 90 days prior to enrollment in this study.
7. Acute illness, including taking antibiotics, analgesics, antipyretics and/or cold medications less than 7 days prior to enrollment in this study.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
NAF cytological classification(s), according to the modified King Classification. | 1 day (single time point)

SECONDARY OUTCOMES:
The IBIS (Tyrer-Cuzick) risk score (10-year and lifetime breast cancer risk estimate. | 1 day (single time point)
Safety, as reported by adverse events experienced after NAF collection with ForeCYTE Breast Aspirator | 1 day (single time point)
micro-RNA (subgroup analysis of BRCA mutation carriers only) | 1 day (single time point)
  development of micro-RNA panel that signals the transition to breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Kylstra, Study Director — Atossa Therapeutics, Inc.
Locations (2):
- Israel (2):
  - The BARUCH PADEH Medical Center, Poria – Neve Oved, Lower Galilee
  - Ziv Medical Center, Safed, Upper Galilee